CLINICAL TRIAL: NCT06639763
Title: Erectile Aid Use in Post-phalloplasty and Post-metoidioplasty Transgender Patients: an Epidemiological Survey
Brief Title: Erectile Aid Use in Post-phalloplasty and Post-metoidioplasty Transgender Patients
Acronym: AID
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0606
Record Dates: First submitted 2024-08-19; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Transgenderism; Erectile Dysfunction; Gender Dysphoria; Sexual Dysfunction
Keywords: Gender dysphoria; Transgender; Phalloplasty; Metoidioplasty; Erectile dysfunction; Sexual function; Genital reconstruction; Reconstructive urology; Erectile aid; Patient Reported Outcome Measures (PROMs); Erection prosthesis; Penile epithesis
MeSH Terms: conditions — Transsexualism; Erectile Dysfunction; Gender Dysphoria; Sexual Dysfunction, Physiological | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Questionnaire — Questionnaire containing a combination of basic epidemiological questions, questions regarding recent sexual activity, questions regarding sexual preference and sexual activity, questions regarding the use of different types of erectile aids, questions regarding satisfaction with the use of these different erectile aid and questions regarding the satisfaction with sexual functioning and the partner relation. Al patients at least 6 months after primary genital gender-affirming surgery and who are sexually active are eligible.

SUMMARY:
This study seeks to explore the various methods used by transgender men for sexual intercourse following phalloplasty or metoidioplasty, focusing on their satisfaction with different erectile aids, as well as the satisfaction of their partners. Phalloplasty and metoidioplasty are gender-affirming surgeries that often require additional aids to achieve the desired sexual function, particularly for penetration. While internal erectile prostheses are common after phalloplasty, they come with high complication rates, leading some patients to opt for non-surgical aids. However, the effectiveness and comfort of these aids are not well-documented. This study aims to fill this gap by examining the types of aids transgender men use, how well these aids meet their sexual needs, and how satisfied both they and their partners are with the outcomes, providing much-needed insight for healthcare providers and patients alike.

DETAILED DESCRIPTION:
Gender dysphoria (GD) is defined as a "marked incongruence between an individuals' experienced or expressed gender and the one they were assigned to at birth". This definition is in accordance with the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Many GD individuals seek medical aid in the form of psychological counseling, hormonal treatment, and, if desired, surgery to align their physical appearance with the perceived gender identity. A part of this population will eventually undergo genital gender affirming surgery (GGAS) to align the appearance of the external genitalia as well. In transgender men, GGAS can be performed as metoidioplasty or phalloplasty with or without the removal of the native external genitalia. In phalloplasty, anatomically sized external genitalia (penis with or without urethra, scrotum, and perineum) are created using on the one hand a donor skin flap (usually from the forearm, upper leg or inguinal region), and on the other hand tissues from the original genitals. In metoidioplasty, the goal is to create anatomically looking but undersized external genitalia in which the clitoris forms the base of a micro-penis. One study in the United States reported that about 3% of transgender men have undergone a phalloplasty and 19% would like to undergo the procedure in the future. For a metoidioplasty, the numbers are 2% and 25%, respectively. One of the reasons for undergoing masculinizing GGAS is to gain the ability to penetrate a partner during intercourse. As there is no erectile tissue present in the neophallus after phalloplasty, penetration is usually not possible without the use of external or internal erectile aids. In metoidioplasty, the phallus does possess erectile tissue but the eventual size of this microphallus is largely dependent on the individually obtained clitoral hypertrophy after hormonal therapy and the body constitution. Therefore, the ability to penetrate a sexual partner after metoidioplasty cannot be assured.

In patients having undergone phalloplasty a multitude of methods for obtaining phallic rigidity are available. One option can be the implantation of an internal erectile prosthesis. These form the main method of attaining penile rigidity after phalloplasty to date. While a multitude of both malleable and inflatable devices are available, these procedures, just as primary GGAS, carry a high risk of complication. Previous research with prostheses originally designed for cisgender men has shown that up to 22% of prostheses was explanted for various reasons including infection, erosion and malfunction within 20 months. Another study showed that only 62% of patients still had their prosthesis in place after 4 years. More recent publications with a prosthesis specifically designed for phalloplasty patients (ZSI TM 475 FtM, Zephyr Surgical Implants, Switzerland, Europe) have shown explantation rates of 19% and 23% at 9 and 18 months respectively. The lack of reliable, and durable erectile devices leads to the fact that a large proportion of patients either chooses for phalloplasty but never goes on the placement of an erectile prothesis or completely abandons the idea of GGAS under the form of phalloplasty at this point in time. As underlined in a recent qualitative study, transgender men may very well be concerned about the complication rates and likely need for additional surgeries associated with the surgical treatments they seek to diminish their gender dysphoria, specifically in penile implant surgery. In addition to internal devices, external ways of obtaining phallic rigidity have been put forward. The use of one or multiple tight condoms with or without the use of self-adhesive bandages tapering the phallus has been reported, as well as the use of penile sleeves readily available on the market or made to measure. Finally, the use of penile lifters or splints has been evaluated in post-phalloplasty individuals with varying results. However, it is unclear which of these erectile aids are most commonly used and, evenly important, how satisfied patients and their partners are with them.

In metoidioplasty, the neophallus does contain cavernosal bodies. However, according to a study in Belgrade in which 813 metoidioplasties were performed, penetration is not possible due to the small size of the neophallus for those who reported sexual intercourse. Other studies report patients who were able to penetrate after metoidioplasty. According to a review by Frey et al. 51% were able to penetrate. Cohanzad et al. reported a technique, extensive metoidioplasty which they performed on 10 people after which 70% were able to obtain an erection rigid enough for penetration. In another study, they used a penile traction device in 10 transgender and 4 cisgender men to increase the length of the phallus after extensive metoidioplasty. The result was a mean penile length increase of 28.42 mm (21-47 ± 6.86). 9 of 11 participants were eventually able to penetrate during sexual intercourse (1 child and 2 virgin singles who had never had sexual contact were excluded). However, it is not stated whether the participants were already capable of penetration before they started using the device. As in cisgender men with erectile dysfunction, some individuals have reported the use of phospho-diesterase 5 inhibitors (PDE5i's) such as Sildenafil or Tadalafil to increase their natural erection. These PDE5i's increase the inflow of blood into the phallus by relaxing the smooth muscle cells in the cavernosal tissue. Another option is intracavernosal injections (ICI's) with Alprostadil. However, knowledge about these two options in post-metoidioplasty individuals is limited. A study by Khorrami et al. examined sexual aspects that are deemed important to those who underwent metoidioplasty. They found that being able to get and maintain an erection was very important in up to 93% of studied individuals, but only 40% valued the ability to have penetrative intercourse equally. An explanation would be because patients do not expect to get a phallus large enough for penetration after metoidioplasty. Thus, the reason they use PDE5i or ICI to improve erection is not only to penetrate the partner, but also because a better erection allegedly also makes for a better orgasm. Another study by Neuville et al. describes the possibility of a semi-rigid prosthesis for metoidioplasty. This technique seems to be successful in terms of post-operative satisfaction, regrets about the surgery and urinary position. However, it is not examined whether penetration during sexual activity with this semi-rigid prosthesis has improved. Other erectile aids used in metoidioplasty apart from PDE5i and ICI are rarely studied.

Apart from the study of Boskey et al., the success and satisfaction rates of these non- surgical erectile aids are unknown or limited to anecdotal reports of individual patients. The erectile aid examined in this study is the Elator. This device seems to be a good option for penetrative sex in trans men who do not (yet) want an internal prosthesis. However, the results showed that only a few couples were able to use the device effectively to have intercourse in the way they envisioned beforehand. For the majority of the studied population, the Elator proved uncomfortable during use, or did not appear to have the right fit since the device was originally designed for cis-men and the phallus of transmen has a different anatomy. A limitation of this study, however, is the small study population.

Given that no prescription or medical intervention is required to obtain these non-surgical aids, only a small portion of the population that does not opt for an internal prosthesis is still on the physician's radar. The limited knowledge on erectile aids in scientific literature makes it difficult for health care providers to offer supported advice to post-surgical transgender individuals in search of alternatives to surgically implanted erection prostheses.

The purpose of this study is to investigate what methods are used for sexual intercourse by transgender men who have undergone phalloplasty or metoidioplasty and how satisfied they and their partners are with these erectile aids. All patients who are sexually active and at least 6 months after primary genital gender-affirming surgery are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Patient and partner age ≥ 18 years.
* Transgender or gender non-conforming individuals (and their partners).
* Patients have undergone phalloplasty or metoidioplasty as a form of genital gender affirming surgery.
* ≥6 months after phalloplasty or metoidioplasty (any type of flap or technique is allowed).
* Sexually active or has been sexually active since phalloplasty or metoidioplasty with a partner or main sexual partner.
* Voluntarily agreed that the data may be used for an anonymized scientific study.

Exclusion Criteria:

* Patient age < 18 years.
* Cisgender patients treated with phalloplasty or metoidioplasty for various reasons.
* <6 months after phalloplasty or metoidioplasty.
* Not sexually active since phalloplasty/metoidioplasty.
* Patient and/or partner have no interest in penetrative sexual intercourse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Transgender male individuals having undergone masculinizing genital gender affirming surgery at least six months ago and who are currently sexually active and are seeking sexual penetration are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-06 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Types of erectile aids used | One time questionnaire at least six months after primary genital gender affirming phalloplasty or metoidioplasty
  A series of closed and open-ended questions are asked meant to uncover what erectile aids are used by post-phalloplasty and post-metoidioplasty individuals and their partners.
Treatment satisfaction | One time questionnaire at least six months after primary genital gender affirming phalloplasty or metoidioplasty
  Assessed using Erectile Dysfunction Inventory of Treatment Satisfaction questionnaire (EDITS).
  The EDITS questionnaire provides two summative scores of 0-44 and 0-20 for patient and partner scores respectively. A higher score indicates a better treatment satisfaction. Higher scores indicate better outcome.

SECONDARY OUTCOMES:
Epidemiology | One time questionnaire at least six months after primary genital gender affirming phalloplasty or metoidioplasty
  Baseline questions regarding speaking language, gender and current anatomy
Quality of sexual experience | One time questionnaire at least six months after primary genital gender affirming phalloplasty or metoidioplasty
  Assessed using Quality of Sexual Experience questionnaire (QSE). The QSE questionnaire provides a summative score between 7 and 49. A higher score indicates a better sexual experience.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Françoise Spinoit, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Department of Urology, University Hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No